CLINICAL TRIAL: NCT00719875
Title: A Dose-escalating and Phase II Clinical Trial of the Histone Deacetylase (HDAC) Inhibitor Vorinostat (Suberoylanilide Hydroxamic Acid, SAHA, ZolinzaTM) in Combination With Capecitabine (XelodaTM) Using a New Weekly Dose Regimen for Advanced Breast Cancer
Brief Title: HDAC Inhibitor Vorinostat (SAHA) With Capecitabine (Xeloda) Using a New Weekly Dose Regimen for Advanced Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0803003591
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Vorinostat; Histone Deacetylase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Vorinostat

INTERVENTIONS:
Drug: Vorinostat — BID days -7, 1-7 and 15-21, 200 mg
  Other Names: SAHA; Zolinza; HDAC inhibitor; suberoylanilide hydroxamic acid

SUMMARY:
The purpose of this study is to determine the safety profile, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), of oral vorinostat in combination with oral capecitabine given on days 1-7 and 15-21 of a 28 day cycle in patients with advanced breast cancer, using RECIST criteria.

This study was originally intended to be a phase 1/phase 2. The protocol was amended to make this study a phase 1 only.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced breast cancer
* For the dose escalation phase: Patients must be refractory to standard therapy or for which no curative standard therapy exists, to be considered.
* For the phase II: Patients with histologically confirmed metastatic breast cancer who have had no more than 2 prior chemotherapy regimens for treatment of their metastatic breast cancer.
* Metastatic disease should not be progressing so as to require palliative treatment within 4 weeks of enrollment based on clinical assessment by the investigator.
* Development of new lesions or an increase in preexisting lesions on bone scintigraphy, CT, MRI or by physical examination. Patients in whom the sole criterion for progression is an increase in a biochemical marker, e.g., carcinoembryonic antigen (CEA), or an increase in symptoms, are not eligible.
* No radiotherapy, treatment with cytotoxic agents, or treatment with biologic agents within the 4 weeks prior to beginning treatment on this study (6 weeks for mitomycin or nitrosoureas). At least 2 weeks must have elapsed from any prior surgery or hormonal therapy. Patients must have fully recovered from the acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤ grade 1 are eligible.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Life expectancy of greater than 3 months
* Patients must have normal organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m² for patients with creatinine levels above institutional normal.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or capecitabine.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women that are pregnant or breast-feeding are excluded from this study.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and the potential pharmacokinetic interaction between antiretroviral therapy and the investigational agents.
* Patient had prior treatment with an HDAC inhibitor. Patients who have received compounds with HDAC inhibitor-like activity, such as valproic acid, as anti-tumor therapy should not enroll in this study. Patients who have received such compounds for other indications, e.g. valproic acid for epilepsy, may enroll after a 30-day washout period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To determine the safety, dose-limiting toxicities and maximum tolerated dose of oral capecitabine in combination with oral vorinostat given twice a day and to determine the objective response rate using RECIST criteria | Upon completion of study

SECONDARY OUTCOMES:
To determine the clinical benefit, time to progression, and duration of response, in patients with metastatic breast cancer treated with this combination | Upon completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-Khalaf, M.D., Principal Investigator — Yale Unviversity School of Medicine
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States